CLINICAL TRIAL: NCT02748473
Title: Effectiveness of Adding Voluntary Pelvic Floor Muscle Contraction to a Pilates Exercises Program: An Assessor-masked Randomized Controlled Trial
Brief Title: Effectiveness of Adding Voluntary Pelvic Floor Muscle Contraction to a Pilates Exercises Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Luiza Torelli de Souza, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LTS-001
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Sedentary Lifestyle
Keywords: Pilates exercises; pelvic floor muscle contraction
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- pelvic floor muscle strength (Other): evaluated pelvic floor muscle strength before and after Pilates exercises program on sedentary nulliparous women
  Interventions: Other: Pilates Exercises program; Other: Pelvic floor muscle strength; Other: 3D perineal ultrasound
- Device: 3D perineal ultrasound (Other): evaluated the pubovisceral muscle thickness and the levator hiatus area before and after Pilates exercises program on sedentary nulliparous women
  Interventions: Other: Pilates Exercises program; Other: 3D perineal ultrasound

INTERVENTIONS:
Other: Pilates Exercises program — The volunteers were divided in two groups:
  Group I: Pilates exercise program involving only the Pilates exercises protocol Group II: Pilates exercises program with voluntary pelvic floor muscle contraction.
  The protocol of both groups consisted of 24 bi-weekly 1-h individual sessions of Pilates exercises program.
  Both groups performed the same protocol . For the group PEP + PFMC the instructor asked for the maximum contraction muscle of the pelvic floor muscle, during expirations with 5 repetitions performed alternately, thus avoiding pelvic floor muscle exhaustion.
  After the 24 sessions, both groups were retested with the same measured methods of the baseline.
Other: Pelvic floor muscle strength — evaluated the pelvic floor strength by oxford scale and vaginal pressure before and after the 12 sessions with Pilates Exercises Program on sedentary nulliparous women
  Arms: pelvic floor muscle strength
Other: 3D perineal ultrasound — evaluated the pubovisceral muscle thickness and levator hiatus area by 3D perineal ultrasound before and after the 12 sessions with Pilates Exercises Program on sedentary nulliparous women

SUMMARY:
Adding voluntary pelvic floor muscle contraction to a Pilates exercises program can improve the pelvic floor muscle strength on sedentary nulliparous women.

DETAILED DESCRIPTION:
Introduction: The purpose of this study was to evaluate the effectiveness of adding voluntary pelvic floor muscle contraction (PFMC) contraction to a Pilates exercise program on sedentary nulliparous women.

Methods: Fifty-seven healthy nulliparous and physically inactive women were randomized to Pilates exercise program (PEP) with or without PFMC. Forty-eight women concluded this study (24 participants for each group). Every women evaluated before and after the PEP, by a one physiotherapist and an urogynecologist (UG). Both professionals were not revealed to them. This physiotherapist measured their pelvic floor muscle strength by using both, a perineometer (Peritron) and vaginal palpation (Oxford Scale) . The UG, who performed 3D perineal ultrasound exams, collected their data and evaluated the results for pubovisceral muscle thickness and the levator hiatus (LA) area. Both professional were masked to the group allocation. The protocol for both groups consisted of 24 bi-weekly 1-h individual sessions of Pilates exercises, developed by another physiotherapist who is specialized in PFM rehabilitation and Pilates technique.

Group I: Pilates exercise program (PEP), involving only the Pilates exercises protocol without any instruction of a voluntary pelvic floor muscle contraction. I other words, the researcher had, under no circumstance, never explained anything about a voluntary pelvic floor muscle contraction during the Pilates exercise performance.

Group II: Pilates exercises program with voluntary pelvic floor muscle contraction (PEP+PFMC) composed of a Pilates exercises program with voluntary pelvic floor contractions. This included maximum contraction of the pelvic floor muscles during expiratory period with 5 repetitions alternately, thus avoiding any muscle exhaustion pelvic floor that could happen.

ELIGIBILITY:
Inclusion Criteria:

* healthy women (without any gynecologic/neurologic disease)
* sedentary women (do not practice regularly physical activities)
* nulliparous,
* on reproductive age
* with no history of pelvic floor disorders
* capable to perform correct PFMC.

Exclusion Criteria:

* Women were not included if they were not able to perform a correct PFMC.
* Potential subjects were excluded if they had chronic degenerative diseases affecting muscular and nerve tissues, diabetes, cerebrovascular disease or overt neurological conditions,
* pregnancy,
* autoimmune connective tissue disorders
* had previously undergone pelvic floor re-education programs and/or pelvic floor surgery.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
change in Oxford Scale | baseline and 3 months
  evaluated the oxford scale

SECONDARY OUTCOMES:
change in pubovisceral muscle thickness | baseline and 3 months
  evaluated the pubovisceral muscle thickness
change in levator hiatus area | baseline and 3 months
  evaluated the levator hiatus area
change in vaginal pressure | baseline and 3 months
  evaluated the vaginal pressure ( perineometer)

IPD SHARING:
Plan to Share IPD: Undecided